CLINICAL TRIAL: NCT04278677
Title: Sleep Quality and Pain Medication Use Following Arthroscopic Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020 TJ 02
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: This is a provider-crossover study design.
Who Masked: Participant
Masking Description: This is a provider-crossover study design: subjects will receive treatment according to their provider's standard of care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin supplementation (Active Comparator): 5mg melatonin tablets to be taken for 6 weeks
  Interventions: Dietary Supplement: melatonin
- No supplementation (No Intervention)

INTERVENTIONS:
Dietary Supplement: melatonin — Melatonin capsules to be taken for 6 weeks
  Arms: Melatonin supplementation

SUMMARY:
The purpose of this study is to investigate if oral melatonin reduces postoperative sleep 18 disturbances and narcotics use. We will enroll patients undergoing primary arthroscopic rotator 19 cuff repair (ARCR) at the Rothman Institute.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo primary ARCR
* Patient willing and able to complete postoperative surveys

Exclusion Criteria:

* Daily melatonin use for > 1 week during the last 3 months
* Irreparable tears
* Revision rotator cuff repairs
* Severe glenohumeral arthritis
* Concurrent adhesive capsulitis
* Age less than 18
* Pregnancy
* History of substance abuse (drug or alcohol)
* Workman's comp patient or patient has current litigation pending
* Allergy to melatonin
* History of delirium/psychiatric/depression/ on antidepressants
* History of insomnia/ on sleep aid medication
* Use of prescription sedatives
* use of Zelboraf (vemurafenib)
* Use of all blood thinning medications besides aspirin (warfarin, plavix, lovenox, etc.)
* Sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | 6 weeks post-surgery
  PSQI is a validated outcome measure for sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedics at Egg Harbor Township, Egg Harbor, New Jersey, United States

REFERENCES:
- [Derived] Perez AR, Destine H, Patel NK, Campbell RE, Muchintala R, Hall AT, Pepe MD, Tucker BS, Tjoumakaris FP. Effects of Melatonin on Sleep Quality and Patient-Reported Outcomes After Arthroscopic Rotator Cuff Surgery: A Prospective Randomized Controlled Trial. Am J Sports Med. 2024 Oct;52(12):3075-3083. doi: 10.1177/03635465241272076. Epub 2024 Sep 15. PMID 39279257